CLINICAL TRIAL: NCT04406948
Title: Randomized, Double Blind, Placebo Controlled, Parallel Design Phase II b Study of Safety and Efficacy of MGCND00EP1 as an Add on Treatment in Children and Adolescents With Resistant Epilepsies
Brief Title: Study of Safety and Efficacy of MGCND00EP1 as an Add on Treatment in Children and Adolescents With Resistant Epilepsies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to overcome bureaucratic obstacles within timeframe.
Sponsor: MGC Pharmaceuticals d.o.o (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGC-002
Record Dates: First submitted 2020-05-17; First posted 2020-05-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Resistant Epilepsy, Drug; Adolescent Epilepsy; Children Epilepsy; Children and Adolescents With Resistant Epilepsies
Keywords: epilepsy; resistant epilepsy; adolescents; children
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — nabiximols; Electrocardiography; Electroencephalography; Blood Specimen Collection; Urine Specimen Collection; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: * Treatment with current antiepileptic therapy 28 days - Various combinations of anti-epileptic (AE) medications
  * Add on treatment 42 days (6 weeks) - titration period - MGCND00EP1 or placebo in addition to AE medications.
  * Add on treatment 42 days (6 weeks) Maintenance stable treatment period - MGCND00EP1 or placebo in addition to AE medications
  * Add on treatment 14 days (2 weeks)- taper - down titration period - MGCND00EP1 or placebo in addition to AE medications
  * Follow up 28 days - Standard/ previous AE treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGCND00EP1 (Experimental): Participants who will assigned to receive add on MGCND00EP1 will receive carrier oil containing THC and CBD in ratio 20:1, (10% of cannabidiol and 0.5 % and (-)-trans-Δ9-tetrahydrocannabinol) .
  Titration Dose: 1 to 2 mg/kg body weight/day. dose will be increased every week by 2 mg/kg body weight/day up to a maximum 25 mg/kg body weigh/day or maximum daily dose 800 mg (the smaller of those 2 values) (divided into two daily doses).
  After titration, patients will be receiving a stable maintenance dose of IMP (up to 25 mg/kg BW per day or maximum daily dose 800 mg (whichever smaller)) for 6 weeks period.
  During forth treatment period participants will commence a 2 weeks down-titration taper period, followed by 4 weeks observational follow up period of previous standard AE treatment without IMP.
  Interventions: Drug: MGCND00EP1; Diagnostic Test: ECG; Diagnostic Test: EEG; Diagnostic Test: Blood and urine collection
- PLACEBO (Placebo Comparator): Participants who are assigned to receive add on PLACEBO will be administered the carrier oil (without the active ingredients).
  Titration Dose: 1 to 2 mg/kg body weight/day. dose will be increased every week by 2 mg/kg body weight/day up to a maximum 25 mg/kg body weigh/day or maximum daily dose 800 mg (the smaller of those 2 values) (divided into two daily doses).
  After titration, patients will be receiving a stable maintenance dose of IMP (up to 25 mg/kg BW per day or maximum daily dose 800 mg (whichever smaller)) for 6 weeks period.
  During forth treatment period participants will commence a 2 weeks down-titration taper period, followed by 4 weeks observational follow up period of previous standard AE treatment without IMP.
  Interventions: Drug: Placebo; Diagnostic Test: ECG; Diagnostic Test: EEG; Diagnostic Test: Blood and urine collection

INTERVENTIONS:
Drug: MGCND00EP1 — Patients will take cannabis oil during the study
  Other Names: Cannabis oil
  Arms: MGCND00EP1
Drug: Placebo — Patient will take carrier oil during the study
  Arms: PLACEBO
Diagnostic Test: ECG — A standard 12-lead ECG will be recorded using digital ECG recording equipment provided to the investigational site. The ECG has to be performed prior to laboratory samplings at time points indicated in the Schedule of Assessments.
  The ECG recording will be reviewed by investigator and case of need consultation with cardiologist will be performed. The investigator has the final decision on the clinical significance of the ECG results.
Diagnostic Test: EEG — An EEG is an electrophysiological monitoring method that records the electrical activity and measures voltage fluctuations resulting from ionic current within the neurons of the brain. In clinical contexts, EEG refers to the recording of the brain's spontaneous electrical activity over a period of time.
Diagnostic Test: Blood and urine collection — safety blood tests - hematology\blood count and biochemistry standard blood tests urinalysis - urine test analysis
  Other Names: blood tests

SUMMARY:
EudraCT: 2018-003887-29

Objective:To evaluate the safety and efficacy of: MGCND00EP1 from MGC PHARMACEUTICALS d.o.o.

Study Design: Randomized, double blind, placebo controlled parallel grouped study Sample Size: 103 subjects Study Population: Children from 1 year to 18 years of age Comparator Product :Placebo solution, oral IMP Product : MGCND00EP1 (each ml of solution containing 100 mg of cannabidiol and 5 mg of (-)-trans-Δ9- tetrahydrocannabinol as active substance) from MGC PHARMACEUTICALS D.O.O.

According to dosing scheme up to 25 mg/kg BW per day or maximum daily dose 800 mg (whichever smaller) for 6 weeks titration and 6 weeks of treatment, oral administration

DETAILED DESCRIPTION:
Subjects on regular therapy with anti-epileptic medications who have evidence from clinical monitoring that current therapy is insufficient, following failure of at least two AEDs for at least during the last 2 months will be enrolled into this study. Upon subjects/parents have consented to participation in the study and after baseline examinations, subjects will continue with current antiepileptic treatment, as clinically needed, for another 28 days at the same dose as before entering the study; drug accountability will be performed for verification of treatment compliance, and diary will be used to record data on epileptic seizures. After that, participating patients will be randomly assigned to MGCND00EP1 or placebo and take it as add on to previous treatment for 6 weeks as titration period and 6 weeks at maintenance dose, and then titrated down during next two weeks. Patients will continue previous anti- epileptic treatment throughout all the periods of the study.

Day one - Screening and Enrollment Visit :

Total 103 patients: Obtain informed consent from legal guardian. Screen potential subjects by inclusion and exclusion criteria. Visit 1: obtain medical and medication history, vital signs, physical and neurological exam, blood and urine tests, ECG, EEG, concomitant medications, questionnaires.

Weeks 1-4 - AED Stabilization Period :

Visit 2: vital signs, weight, physical and neurological exam, blood and urine tests, concomitant medications, questionnaires, monitor AEs, PK blood collection (subset of patients), randomize and dispense study drugs

Patients will be randomized and will either get placebo or MGCND00EP1 (3:1 active:placebo)

Weeks 5-10 - Dose titration period:

Dose escalations (2 mg/kg body weight/day increments), as required, up to 25 mg/kg/day or 800 mg/day, the lower of the two, until stable dose is reached.

Visit 3: vital signs, weight, physical and neurological exam, blood and urine tests, concomitant medications, questionnaires, collect and issue diaries, dispense study drug, monitor AEs

Weeks 11-16 - Maintenance Period :

Visit 4: vital signs,weight, physical and neurological exam, blood and urine tests, concomitant medications, questionnaires, PK sample collection (subset of patients), collect and issue diaries, dispense study drug, EEG, monitor AEs

Weeks 17-18 - Tapering-off and Follow-up Period:

Weekly phone call to determine taper dose at physician's discretion

Visit 5: vital signs,weight, physical and neurological exam, blood and urine tests, concomitant medications, questionnaires, monitor AEs, collect diaries and unused drug

Weeks 19-20 - Follow-up Period:

Weekly phone calls

Visits 6: vital signs,weight, physical and neurological exam, concomitant medications, monitor AEs, collect diaries .

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented clinically confirmed diagnosis of epilepsy;
* Patient did not respond to at least 2 AED's therapy given in adequate doses;
* Patients current therapy is considered inadequate (not completely controlled by AEDs); patients had four or more countable seizures with a motor component per 4 week period;
* Patient is aged 1 year - 18 years inclusive at screening age;
* Patient took one or more AEDs treatment at dose which has been stable for at least 4 weeks before enrolment;
* Females of childbearing potential can only participate in the study if willing to use acceptable, effective methods of contraception during the trial and for three month after end of trial participation as defined in point 7.10 of this protocol;
* Patient/parent is able to read/understand informed consent.
* Male patients must either be surgically sterile or he and his female spouse/partner who is of childbearing potential must be willing to use highly effective methods of contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the study.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation (VNS) were stable for four weeks prior to screening and participants were willing to maintain a stable regimen throughout the study. The ketogenic diet and VNS treatments are not counted as an AED.

Exclusion Criteria:

* Known history or presence of clinically significant unstable medical condition other that epilepsy which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Known history or presence of serious cardiovascular disease
* Known or suspected history or family history of: schizophrenia, or other psychotic illness, severe personality disorder or other significant psychiatric disorder.
* Known or suspected allergy hypersensitivity or idiosyncratic reaction to cannabinoids or any other drug substances with similar activity or to any of the excipients of the IMP.
* Participant has clinically relevant abnormalities in the 12-lead electrocardiogram measured at screening or randomisation.
* Patients were currently using or had in the past used recreational or medicinal cannabis or synthetic CBD based medications or preparations within last 3 months or had previous or current treatment with cannabis-based therapy within last 3 months.
* History of drug or alcohol addiction requiring treatment.
* History of malabsorption within the last year or presence of clinically significant gastrointestinal disease or surgery that may affect drug bioavailability, including but not limited to cholecystectomy.
* Presence of hepatic or renal dysfunction.
* Females who: are pregnant (serum hCG level consistent with pregnancy diagnosis); or are lactating;
* Participation in a clinical trial that involved administration of an investigational medicinal product within 90 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results;
* Participant has clinically significant abnormal laboratory values (e.g. liver enzymes);
* Participant has clinically significant findings from a physical examination (fever);
* In case of ketogenic diet or VNS; the diet need to be stable for at least 4 weeks, and VNS ramping needs to be stable at least 12 weeks before enrolment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients showing a >50% reduction in frequency of seizures at week 12 of the study, in the treatment versus placebo groups | 12 weeks
  study drug overall efficiency as a seizure reducing treatment compared to placebo group
Change in number of epileptic seizures as documented by patient diaries (Visit 2 level compared to Visit 3 level and Visit 4) in treatment and placebo group. | 16 weeks
  study drug overall efficiency as a seizure reducing treatment

SECONDARY OUTCOMES:
The incidence of adverse events will be summarized by organ class, severity and duration on weeks 12 and 18 of the study. | 12-18 weeks
  Adverse events assessment
Any change in physical examination, vital signs, lab tests results, ect will be collected and analyzed. | 18 weeks
  Improvement in vital signs, lab test results and physical examination
Change in duration of epileptic seizures as documented by patient diaries (Visit 2 level compared to Visit 3 level and Visit 4 level compared to Visit 2 level) by treatment group. | 12-18 weeks
  seizure frequency assessment
Change in score from Quality of Life in Childhood Epilepsy Questionnaire 55 (QOLCE-55 questionnaire) scoring 0-100 points, higher scoring indicates better condition. scoring will be compared between Visit 2 level and Visit 4 level. | 18 weeks
  QoL questionnaire assessment
Change in Clinical Global Impressions Scale (CGI scale) scoring 1-7 points, low scoring indicates better condition. Visit 2 level compared to Visit 4 level by treatment group. | 18 weeks
  CGI improvement by treatment group
Percentage of MGCND00EP1-treated patients who will develop a response to MGCND00EP1 (response will be defined as a reduction of seizures frequency by at least 25 % ) as compared between Visit 2 level and Visit 4 level | 18 weeks
  response to MGCND00EP1
Proportion of seizure-free patients between the placebo and treatment group on week 12 of treatment (including titration). | 12 weeks
  Proportion of seizure-free patients
Change in form of new seizures and emergency of new forms will be monitored during the trial | 18 weeks
  New seizure or seizure form emergency

CONTACTS AND LOCATIONS:
Overall Officials: Rubi Zomer, Study Director — MGC Pharmacuticals
Locations (2):
- Schneider Children's Medical Center of Israel, Petach Tikvah, Central District, Israel
- University Children's Hospital Ljubljana University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg AT, Zelko FA, Levy SR, Testa FM. Age at onset of epilepsy, pharmacoresistance, and cognitive outcomes: a prospective cohort study. Neurology. 2012 Sep 25;79(13):1384-91. doi: 10.1212/WNL.0b013e31826c1b55. Epub 2012 Sep 12. PMID 22972641
- [Background] Devinsky O, Vickrey BG, Cramer J, Perrine K, Hermann B, Meador K, Hays RD. Development of the quality of life in epilepsy inventory. Epilepsia. 1995 Nov;36(11):1089-104. doi: 10.1111/j.1528-1157.1995.tb00467.x. PMID 7588453
- [Background] Donner EJ. Opportunity gained, opportunity lost: treating pharmacoresistant epilepsy in children. Epilepsia. 2013 May;54 Suppl 2:16-8. doi: 10.1111/epi.12178. PMID 23646965
- [Background] Cilio MR, Thiele EA, Devinsky O. The case for assessing cannabidiol in epilepsy. Epilepsia. 2014 Jun;55(6):787-90. doi: 10.1111/epi.12635. Epub 2014 May 22. PMID 24854434
- [Background] Maa E, Figi P. The case for medical marijuana in epilepsy. Epilepsia. 2014 Jun;55(6):783-6. doi: 10.1111/epi.12610. Epub 2014 May 22. PMID 24854149
- [Background] Sharp GB, Samanta D, Willis E. Options for pharmacoresistant epilepsy in children: when medications don't work. Pediatr Ann. 2015 Feb;44(2):e43-8. doi: 10.3928/00904481-20150203-11. PMID 25658218
- [Background] Bent S. Herbal medicine in the United States: review of efficacy, safety, and regulation: grand rounds at University of California, San Francisco Medical Center. J Gen Intern Med. 2008 Jun;23(6):854-9. doi: 10.1007/s11606-008-0632-y. Epub 2008 Apr 16. PMID 18415652
- [Background] Russo EB. History of cannabis and its preparations in saga, science, and sobriquet. Chem Biodivers. 2007 Aug;4(8):1614-48. doi: 10.1002/cbdv.200790144. PMID 17712811
- [Background] Zuardi AW, Crippa JA, Hallak JE, Moreira FA, Guimaraes FS. Cannabidiol, a Cannabis sativa constituent, as an antipsychotic drug. Braz J Med Biol Res. 2006 Apr;39(4):421-9. doi: 10.1590/s0100-879x2006000400001. Epub 2006 Apr 3. PMID 16612464
- [Background] Devinsky O, Marsh E, Friedman D, Thiele E, Laux L, Sullivan J, Miller I, Flamini R, Wilfong A, Filloux F, Wong M, Tilton N, Bruno P, Bluvstein J, Hedlund J, Kamens R, Maclean J, Nangia S, Singhal NS, Wilson CA, Patel A, Cilio MR. Cannabidiol in patients with treatment-resistant epilepsy: an open-label interventional trial. Lancet Neurol. 2016 Mar;15(3):270-8. doi: 10.1016/S1474-4422(15)00379-8. Epub 2015 Dec 24. PMID 26724101
- [Background] Cortesi M, Fusar-Poli P. Potential therapeutical effects of cannabidiol in children with pharmacoresistant epilepsy. Med Hypotheses. 2007;68(4):920-1. doi: 10.1016/j.mehy.2006.09.030. Epub 2006 Nov 16. No abstract available. PMID 17112679
- [Background] Dan B. Cannabinoids in paediatric neurology. Dev Med Child Neurol. 2015 Nov;57(11):984. doi: 10.1111/dmcn.12926. No abstract available. PMID 26443475
- [Background] Press CA, Knupp KG, Chapman KE. Parental reporting of response to oral cannabis extracts for treatment of refractory epilepsy. Epilepsy Behav. 2015 Apr;45:49-52. doi: 10.1016/j.yebeh.2015.02.043. Epub 2015 Apr 3. PMID 25845492
- [Background] Devinsky O, Cilio MR, Cross H, Fernandez-Ruiz J, French J, Hill C, Katz R, Di Marzo V, Jutras-Aswad D, Notcutt WG, Martinez-Orgado J, Robson PJ, Rohrback BG, Thiele E, Whalley B, Friedman D. Cannabidiol: pharmacology and potential therapeutic role in epilepsy and other neuropsychiatric disorders. Epilepsia. 2014 Jun;55(6):791-802. doi: 10.1111/epi.12631. Epub 2014 May 22. PMID 24854329
- [Background] Bergamaschi MM, Queiroz RH, Zuardi AW, Crippa JA. Safety and side effects of cannabidiol, a Cannabis sativa constituent. Curr Drug Saf. 2011 Sep 1;6(4):237-49. doi: 10.2174/157488611798280924. PMID 22129319
- [Background] Koppel BS, Brust JC, Fife T, Bronstein J, Youssof S, Gronseth G, Gloss D. Systematic review: efficacy and safety of medical marijuana in selected neurologic disorders [RETIRED]: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Apr 29;82(17):1556-63. doi: 10.1212/WNL.0000000000000363. PMID 24778283
- [Background] Izquierdo I, Tannhauser M. Letter: The effect of cannabidiol on maximal electroshock seizures in rats. J Pharm Pharmacol. 1973 Nov;25(11):916-7. doi: 10.1111/j.2042-7158.1973.tb09976.x. No abstract available. PMID 4149660
- [Background] Chesher GB, Jackson DM, Malor RM. Interaction of delta9-tetrahydrocannabinol and cannabidiol with phenobarbitone in protecting mice from electrically induced convulsions. J Pharm Pharmacol. 1975 Aug;27(8):608-9. doi: 10.1111/j.2042-7158.1975.tb09515.x. No abstract available. PMID 239178
- [Background] Jones NA, Hill AJ, Smith I, Bevan SA, Williams CM, Whalley BJ, Stephens GJ. Cannabidiol displays antiepileptiform and antiseizure properties in vitro and in vivo. J Pharmacol Exp Ther. 2010 Feb;332(2):569-77. doi: 10.1124/jpet.109.159145. Epub 2009 Nov 11. PMID 19906779
- [Background] Mula M. Investigational new drugs for focal epilepsy. Expert Opin Investig Drugs. 2016;25(1):1-5. doi: 10.1517/13543784.2016.1110144. Epub 2015 Nov 4. PMID 26535466
- [Background] Hess EJ, Moody KA, Geffrey AL, Pollack SF, Skirvin LA, Bruno PL, Paolini JL, Thiele EA. Cannabidiol as a new treatment for drug-resistant epilepsy in tuberous sclerosis complex. Epilepsia. 2016 Oct;57(10):1617-1624. doi: 10.1111/epi.13499. Epub 2016 Oct 3. PMID 27696387
- [Background] Tzadok M, Uliel-Siboni S, Linder I, Kramer U, Epstein O, Menascu S, Nissenkorn A, Yosef OB, Hyman E, Granot D, Dor M, Lerman-Sagie T, Ben-Zeev B. CBD-enriched medical cannabis for intractable pediatric epilepsy: The current Israeli experience. Seizure. 2016 Feb;35:41-4. doi: 10.1016/j.seizure.2016.01.004. Epub 2016 Jan 6. PMID 26800377
- [Background] Goldstein B. Cannabis in the treatment of pediatric epilepsy. O'Shaugnessy's 2016:7-9.
- [Background] Reddy DS, Golub VM. The Pharmacological Basis of Cannabis Therapy for Epilepsy. J Pharmacol Exp Ther. 2016 Apr;357(1):45-55. doi: 10.1124/jpet.115.230151. Epub 2016 Jan 19. PMID 26787773
- [Background] Geffrey AL, Pollack SF, Bruno PL, Thiele EA. Drug-drug interaction between clobazam and cannabidiol in children with refractory epilepsy. Epilepsia. 2015 Aug;56(8):1246-51. doi: 10.1111/epi.13060. Epub 2015 Jun 26. PMID 26114620
- [Background] O'Connell BK, Gloss D, Devinsky O. Cannabinoids in treatment-resistant epilepsy: A review. Epilepsy Behav. 2017 May;70(Pt B):341-348. doi: 10.1016/j.yebeh.2016.11.012. Epub 2017 Feb 8. PMID 28188044
- [Background] Goodwin SW, Lambrinos AI, Ferro MA, Sabaz M, Speechley KN. Development and assessment of a shortened Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55). Epilepsia. 2015 Jun;56(6):864-72. doi: 10.1111/epi.13000. Epub 2015 Apr 25. PMID 25912151
- [Background] Conway L, Widjaja E, Smith ML, Speechley KN, Ferro MA. Validating the shortened Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55) in a sample of children with drug-resistant epilepsy. Epilepsia. 2017 Apr;58(4):646-656. doi: 10.1111/epi.13697. Epub 2017 Feb 15. PMID 28199002
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Bornheim LM, Everhart ET, Li J, Correia MA. Induction and genetic regulation of mouse hepatic cytochrome P450 by cannabidiol. Biochem Pharmacol. 1994 Jul 5;48(1):161-71. doi: 10.1016/0006-2952(94)90236-4. PMID 8043019
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Mortati K, Dworetzky B, Devinsky O. Marijuana: an effective antiepileptic treatment in partial epilepsy? A case report and review of the literature. Rev Neurol Dis. 2007 Spring;4(2):103-6. PMID 17609644
- [Background] Volkow ND, Compton WM, Weiss SR. Adverse health effects of marijuana use. N Engl J Med. 2014 Aug 28;371(9):879. doi: 10.1056/NEJMc1407928. No abstract available. PMID 25162899
- [Background] Porter BE, Jacobson C. Report of a parent survey of cannabidiol-enriched cannabis use in pediatric treatment-resistant epilepsy. Epilepsy Behav. 2013 Dec;29(3):574-7. doi: 10.1016/j.yebeh.2013.08.037. PMID 24237632
- [Background] Gloss D, Vickrey B. Cannabinoids for epilepsy. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD009270. doi: 10.1002/14651858.CD009270.pub2. PMID 22696383
- [Background] Zaccara G, Giovannelli F, Schmidt D. Placebo and nocebo responses in drug trials of epilepsy. Epilepsy Behav. 2015 Feb;43:128-34. doi: 10.1016/j.yebeh.2014.12.004. Epub 2015 Feb 19. PMID 25703333
- [Background] Sativex smpc , 20.09.2018
- [Background] Wall ME, Sadler BM, Brine D, Taylor H, Perez-Reyes M. Metabolism, disposition, and kinetics of delta-9-tetrahydrocannabinol in men and women. Clin Pharmacol Ther. 1983 Sep;34(3):352-63. doi: 10.1038/clpt.1983.179. PMID 6309462
- [Background] Ohlsson A, Lindgren JE, Wahlen A, Agurell S, Hollister LE, Gillespie HK. Plasma delta-9 tetrahydrocannabinol concentrations and clinical effects after oral and intravenous administration and smoking. Clin Pharmacol Ther. 1980 Sep;28(3):409-16. doi: 10.1038/clpt.1980.181. PMID 6250760
- See also: nice.org-( dne: 14.februarja 2016) — https://www.nice.org.uk/guidance/cg137/chapter/1-Guidance